CLINICAL TRIAL: NCT03492346
Title: Limb Girdle Muscular Dystrophy Type 2E Recruitment Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Myonexus Therapeutics (Unknown)
Responsible Party: Principal Investigator, Jerry R. Mendell, Principal Investigator, Nationwide Children's Hospital
Other Study IDs: IRB18-00224
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Limb-Girdle Muscular Dystrophy, Type 2E
Keywords: LGMD2E; Limb Girdle Muscular Dystrophy; sarcoglycanopathy; β -sarcoglycan; Natural History
MeSH Terms: conditions — Limb-girdle muscular dystrophy, type 2E; Muscular Dystrophies, Limb-Girdle; Sarcoglycanopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LGMD2E Subject Population: Individuals:
  * Confirmed LGMD2E diagnosis by genetic testing or
  * Suspected of having LGMD type 2E due to symptoms and a diagnosed family member or a member of a community with a large population of one of these two types

SUMMARY:
This study is to recruit and establish baseline measurements for potential subjects that may be eligible for a gene therapy trial. Specifically, this trial is recruiting individuals who are suspected or have been confirmed to have Limb Girdle Muscular Dystrophy type 2E (LGMD2E).

DETAILED DESCRIPTION:
This is a longitudinal observational study. It is a 24-month study with the possibility of extending the data time points. Visits will occur monthly. However, at the discretion of the PI, subjects may not be required to return monthly. These subjects may return at intervals ranging from 2 months to a max of 6 months apart.

In the situation that the subjects would fall out of the inclusion criteria or not be eligible for the LGMD2E gene therapy trial, they will be given the opportunity to roll over into the Natural History for LGMD (IRB17-01086). If a subject is invited to screen for the gene therapy trial they will discontinue this trial. By being in this study, it is not a guarantee that subjects will be invited to screen for the LGMD2E gene therapy trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-15 inclusive
* Males or females of any ethnic group
* SGCB DNA gene mutations at both alleles or suspected to have LGMD2E based on family and medical history. If suspected, genetic testing will be performed to confirm diagnosis.
* Weakness demonstrated based on history of difficulty running, jumping and climbing stairs
* Ability to complete 100MW timed test within 30-90% predicted
* Perform assessments to the best of their ability with reliable results as deemed by the evaluator.
* Ability to attend scheduled appointments
* Ability to provide informed consent (or assent for ages 9-15)

Exclusion Criteria:

* Confirmed diagnosis of neuromuscular disorder other than LGMD2E
* Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with the protocol required testing or procedures or compromise the subject's wellbeing, safety, or clinical interpretability
* Subjects with AAVrh74 binding antibody titers > 1:400 as determined by ELISA immunoassay. If endpoint titer is positive at screening, testing may be repeated in 1 month. Antibody testing will be performed on a separate study (IRB17-01101).
* Diagnosis of (or ongoing treatment for) an autoimmune disease

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * Confirmed LGMD2E diagnosis by genetic testing or
  * Suspected of having LGMD type 2E due to symptoms and a diagnosed family member or a member of a community with a large population of one of these two types
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2023-03-28 (Estimated); Study Completion 2023-03-28 (Estimated)

PRIMARY OUTCOMES:
Baseline Measurements | 2 years
  Establish baseline measurements for potential subjects that may be enrolled into a gene therapy trial.

SECONDARY OUTCOMES:
Disease Progression | 2 years
  Better define the rate of disease progression and skeletal muscle involvement
Registry | 2 years
  Generate a registry of well-characterized LGMD2E patients

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Mendell, M.D., Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States